CLINICAL TRIAL: NCT02774239
Title: A Pilot Trial To Assess The Feasibility And Efficacy Of Subcutaneous Immunoglobulin In Patients With Myasthenia Gravis Exacerbation
Brief Title: A Pilot Trial To Assess The Feasibility And Efficacy Of SCIG In Patients With MG Exacerbation (SCIG-MG)
Acronym: SCIG-MG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZS2013-01
Record Dates: First submitted 2015-04-20; First posted 2016-05-17 (Estimated); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis | interventions — Hizentra

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SC Treatment Period (Experimental): Participants will receive 2gm/kg of Human normal immunoglobulin G (IgG) infused over 4 weeks in a dose escalating manner as follows:
  * 1st week: 2-3 SCIG infusions of 10ml per site at four sites (total dose 16 to 24g)*
  * 2nd week: 2-3 SCIG infusions of 15ml per site at four sites (total dose 24 to 36g)*
  * 3rd week: 2-4 SCIG infusions of 20ml per site at four sites (total dose 32 to 64g)*
  * 4th week: 2-4 SCIG infusions of 25ml per site at four sites (total dose 40 to 80g)*
    * Doses indicated are study recommended. Doses may be adjusted depending on tolerance and total dose required by the patient.
  Interventions: Drug: Human normal immunoglobulin G (IgG)

INTERVENTIONS:
Drug: Human normal immunoglobulin G (IgG) — Study medication is available in the following forms: 5 mL (1 g IgG) in a 5 mL infusion bottle, 10 mL (2 g IgG) in a 10 mL infusion bottle, 20 mL (4 g IgG) in a 20 mL infusion bottle, 50 mL (10 g IgG) in a 50 mL infusion bottle.
  Patients will be receiving 2gm/kg (150gm for a 75kg patient) of 20% SCIG (Hizentra) infused over four weeks in a dose escalating manner.
  Other Names: Hizentra®

SUMMARY:
This is a prospective open-label, uncontrolled, single-blind, pilot clinical trial.

The primary objective is to assess the efficacy, safety, feasibility and tolerability of SCIG in patients with worsening MG.

Participants with moderate worsening of MG symptoms (MGFA Class II and III) who are considered to be appropriate for immunoglobulin therapy will be screened for the study by the treating neurologist.

Patients will be receive 2gm/kg (150gm for a 75kg patient) of 20% SCIG (Hizentra) infused over 4 weeks in a dose escalating manner.

Additionally, this study will be assessing the feasibility of employing SCIG as an alternative therapy to IVIG in patients with MG exacerbation. The cost-effectiveness of SCIG versus IVIG will be evaluated, and the impact of SCIG therapy will be assessed from both a health-resource perspective and from a patient perspective.

DETAILED DESCRIPTION:
This is a prospective open-label, uncontrolled, single-blind, pilot clinical trial.

The primary objective is to assess the efficacy, safety, feasibility and tolerability of SCIG in patients with worsening MG.

Study Rationale and Significance

Subcutaneous immunoglobulin (SCIG) is a novel form of immune therapy for neuromuscular diseases and may offer several advantages over intravenous immunoglobulin (IVIG).

Although no large-scale studies have been in conducted in MG patients, pilot studies with SCIG in multifocal motor neuropathy indicate that it may be a feasible, effective and safe alternative to IVIG in a condition, which like MG, shows excellent response to IVIG infusion.

Patients are able to tolerate it better and have improved quality of life due to added flexibility to the treatment schedule. SCIG is also potentially less expensive than IVIG since the costs associated with inpatient treatment as well as nursing support are saved.

SCIG also has the potential to be more effective and durable since the serum levels of immunoglobulin show a more sustained increase compared to IVIG. A drawback associated with SCIG is the small amount of immunoglobulin that can be infused over a short period. As compared to IVIG where the usual dose (2gm/kg for neuromuscular diseases) can be infused over 2 - 5 days, the same dose of SCIG would require 3 - 4 weeks to be administered with the currently available formulations. This may mean a delayed onset of peak-dose effect and SCIG may not be feasible for MG patients who are rapidly worsening or in MG crisis.

Nevertheless, SCIG may be an attractive option in a large subpopulation of MG patients who have mild to moderate disease exacerbations or who are on maintenance IVIG therapy provided its efficacy, tolerability and feasibility is determined in this patient population.

Methodology

Participants with moderate worsening of MG symptoms (MGFA Class II and III) who are considered to be appropriate for immunoglobulin therapy at the MG clinic at the University of Alberta will be screened for the study by the treating neurologist.

Patients will be receive 2gm/kg (150gm for a 75kg patient) of 20% SCIG (Hizentra) infused over 4 weeks in a dose escalating manner. Participants will undergo infusions two to four times a week, depending on their tolerance, beginning with a dose of 10 ml per site at four injection sites, increasing by 5 ml per week for a total of 25 ml per site at four injection sites after four weeks.

The dose is flexible and will vary based on the patient's tolerance to the medication and the total amount of medication the patient will be receiving based on their body weight. The initial (one or two) doses will be infused within the medical outpatient facility at the University of Alberta Hospital. This will allow for the observation of any infusion reactions and will also serve as nurse-provided self- infusion training sessions for patients.

Participants will be assessed weekly for symptomatic change and reports of satisfaction and quality of life. The primary outcome variable is the change in the Quantitative Myasthenia Gravis (QMG) Score for Disease Severity from baseline to day 42 (6 weeks). A change of 3.5 points will be considered to be clinically significant.

Safety and pharmacokinetic assessments of SCIG will be performed weekly throughout the study.

Additionally, this study will be assessing the feasibility of employing SCIG as an alternative therapy to IVIG in patients with MG exacerbation. The cost-effectiveness of SCIG versus IVIG will be evaluated, and the impact of SCIG therapy will be assessed from both a health-resource perspective and from a patient perspective.

The practicality of using SCIG in patients with MG will be determined by documenting the number of patients who are able to be trained for self- administration of SCIG, and by the patients' self-reported satisfaction with SCIG treatment.

The speed of SCIG treatment onset will also be assessed and compared to IVIG treatment onset. All of these described measures will be used to determine the feasibility and practicality of using SCIG in patients with MG exacerbation and its impact on the healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* Patients between18 to 80 years of age, diagnosed with MG (see below) who have worsening myasthenic symptoms - (defined as increasing diplopia, ptosis, dysarthria, dysphagia, difficulty chewing, or limb weakness severe enough to warrant immunoglobulin therapy.
* MG diagnosis will be based upon the clinical evaluation by a neuromuscular expert and meeting any two of the following supportive criteria:

  1. Abnormal Tensilon test
  2. Abnormal repetitive nerve stimulation studies
  3. Abnormal single fiber electromyography (EMG)
  4. Increased serum acetylcholine receptor or anti-MuSK antibodies
  5. Prior response to immunotherapy

Exclusion Criteria:

1. Respiratory distress requiring ICU admission or a vital capacity <1 L
2. Severe swallowing difficulties with a high risk of aspiration
3. Change in corticosteroid dosage in the 4 weeks prior to screening
4. Known immunoglobulin A (IgA) deficiency
5. Pregnant or breast feeding women
6. Active renal or hepatic insufficiency, clinically significant cardiac disease
7. Patients with worsening weakness associated with an infectious process
8. Previous lack of responsiveness to IVIG
9. History of previous MG crises

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-10; Primary Completion 2022-10-21 (Actual); Study Completion 2022-10-21 (Actual)

PRIMARY OUTCOMES:
Change in Quantitative Myasthenia Gravis Score (QMGS) from baseline to day 42 after treatment. | Baseline - Day 42
  QMGS is a validated clinical measure of myasthenia gravis ranging from 0 points (no myasthenic weakness) to a maximum of 39 points, with a defined change of 3.4 units required for clinical significance.

SECONDARY OUTCOMES:
Quality of life will be assessed through the Quality of Life (QOL) score, a qualitative questionnaire. | Baseline - Day 42
Change in Manual Muscle Testing (MMT) score from baseline to day 42 after treatment. | Baseline - Day 42
  MMT is a validated clinical measure of myasthenia gravis ranging from 0 points (no myasthenic weakness) to a maximum of 128 points, with a defined change of 25% from baseline required for clinical significance.
Adverse events related to SCIG infusions will be recorded if/when they occur. | Baseline - Day 42
Patient satisfaction with the treatment modality will be assessed using a questionnaire. | Day 42
  TQSM: Treatment Satisfaction Questionnaire for Medication. An 11 question ordinal scale measuring responses from "Extremely satisfied" to "Extremely dissatisfied" over a 7 item option list. Questions cover four domains, corresponding to distinct aspects related to the satisfaction of patients with their treatment (Effectiveness; Side effects; Convenience and Global satisfaction). A score can be obtained for each domain by summing of the corresponding items transformed on a 0-100 scale; higher values indicate higher satisfaction, better perceived effectiveness, lower burden associated to side-effects, better convenience
Serious Adverse Events related to SCIG infusions will be recorded if/when they occur. | Baseline - Day 42
Proportion of participants successfully trained will be recorded indicating feasibility based on patient compliance. | Baseline - Week 2
Proportion of participants completing will be recorded indicating feasibility based on patient compliance. | Baseline - Day 42
Myasthenia Gravis (MG) Composite scores will be used to evaluate disease severity through a number of functional assessments, including muscle strength and ability to complete activities of daily living. | Baseline - Day 42

OTHER OUTCOMES:
Cost effectiveness of SCIG therapy will be calculated in comparison to standard IVIG therapy. This will indicate health economics. | Baseline - Day 42
Change in QOL 36 score from Baseline to day 42) | Baseline - Day 42
  Change in Quality of Life (QOL) score from Baseline to day 42.
Time required for the treatments. | Baseline - Day 42
  Average time in minutes required for each infusion session during study. Determined for each participant.
Preference for treatments (Treatment Satisfaction Questionnaire for Medication (TSQM). | Day 42
  11 item scale measuring treatment satisfaction for medication over 3 domains (Effectiveness, Side effects, Convenience, Global Satisfaction). Score from 10 to 43
Intent to continue using SCIG if necessary (Via pt. interview) | Day 42
  Yes= will continue SCIG therapy, No= will not continue SCIG therapy.
Proportion of participants successfully trained in self-administration of SCIG. | Day 2, Day 3.
  Proportion of participants who successfully trained in self-administration of SCIG expressed as a percentage (completed training/underwent training x 100).
Proportion of participants completing the study. | Day 42
  Proportion of patients who completed the study expressed as a percentage (finished study/started study x 100).
Infusion nurse's assessment of this participant population's ability to use this treatment modality (Written impression) | Day 42
  Qualitative measure. Narrative reflecting the infusion nurse's overall impression of target population's ability to employ SCIG within the parameters defined by the study. (data is a written narrative. By definition, this has no units nor is it collected by any instrument (questionnaire, scale parameter ect.) ie. QUALITATIVE data)
Speed of treatment onset of SCIG. | Day 1
  The number of days between prescription of SCIG treatment and infusion of first dose.
Speed of treatment onset of IVIG. | Day 1
  The number of days between prescription of IVIG treatment and infusion of first dose, for any study participant who has received IVIG treatments in the past. This interval will be determined for all available previous IVIG infusions for each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Zaeem A Siddiqi, MD, PhD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - Vancouver General Hospital - Gordon & Leslie Diamond Health Care Centre, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No